CLINICAL TRIAL: NCT02757924
Title: Behavior of Infants Fed a Partially Hydrolyzed Formula Supplemented With Prebiotics
Brief Title: Behavior of Infants Fed Formula Supplemented With Prebiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AL20
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Gastrointestinal Tolerance
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infant formula supplemented with prebiotics (Experimental): infant formula powder, feed ad libitum
  Interventions: Other: Infant formula supplemented with prebiotics

INTERVENTIONS:
Other: Infant formula supplemented with prebiotics — Sole source nutrition

SUMMARY:
To observe the effects of partially hydrolyzed formula supplemented with oligosaccharides on symptoms of formula intolerance in healthy term infants.

ELIGIBILITY:
Inclusion Criteria:

* Subject is judged to be in good health.
* Subject is a singleton from a full-term birth with a gestational age of 37 - 42 weeks.
* Subject's birth weight was ≥ 2490 g (~5 lbs. 8 oz.).
* Infant was identified by parents as very fussy or extremely fussy.
* Infant is exclusively formula-fed at time of study entry. Parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study.
* Parent(s) confirm their intention not to administer vitamin or mineral supplements, solid foods or juices to their infant from enrollment through the duration of the study.

Exclusion Criteria:

* An adverse maternal, fetal or subject medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development.
* Subject is taking and plans to continue medications, home remedies (such as juice for constipation), herbal preparations or rehydration fluids that might affect GI tolerance.
* Subject participates in another study that has not been approved as a concomitant study.
* Subject has been fed any formula containing human milk oligosaccharides prior to study enrollment.
* Subject has been treated with oral antibiotics within 7 days prior to study enrollment.
* Mother intends to use a combination of breast and formula feeding.

Ages: 7 Days to 42 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Fussiness | Change from baseline (3 days prior to study day 1) to within 1 day of initiation of study feeding
  Parent questionnaires

SECONDARY OUTCOMES:
Fussiness | Baseline to Day 29
  Parent Questionnaires
Hours of Daily Crying | Baseline to Day 29
  Parent Questionnaires
Gastrointestinal Tolerance | Baseline to Day 29
  Parent Questionnaires
Stool Pattern | Baseline to Day 29
  Parent Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Borschel, PhD, RD, LD, Study Chair — Abbott Nutrition
Locations (11):
- United States (11):
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Pensacola Research Consultants, Inc, Pensacola, Florida
  - Score Physician Alliance, LLC, St. Petersburg, Florida
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - Aventiv Research, Grove City, Ohio
  - Coastal Pediatric Research, Charleston, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Southwest Children's Research Associates, P.A., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided